CLINICAL TRIAL: NCT04886986
Title: Phase I/II Study of 225Ac-J591 Plus 177Lu-PSMA-I&T for Progressive Metastatic Castration Resistant Prostate Cancer
Brief Title: Phase I/II 225Ac-J591 Plus 177Lu-PSMA-I&T for Progressive Metastatic Castration Resistant Prostate Cancer
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Need to wait until a new collaborator is available and confirmed
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-08022486
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): Patients enrolled in the study will receive the study drugs 225Ac-J591 and 177Lu-PSMA-I&T, along with 68Ga-PSMA-11.
  Interventions: Drug: 225Ac-J591; Drug: 177Lu-PSMA-I&T; Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: 225Ac-J591 — 30 - 40 KBq/kg (dose-escalation) every 8 weeks, for up to 2 cycles. Administered together with 177Lu-PSMA-I&T. Intravenous administration.
Drug: 177Lu-PSMA-I&T — 6.8 GBq (fixed dose) every 8 weeks, for up to 2 cycles. Administered together with 225Ac-J591. Intravenous administration.
  Other Names: 177Lu-PNT2002
Drug: 68Ga-PSMA-11 — [185 ±74 MBq or 5 ±2 mCi] intravenous during screening, 12 weeks, 24 weeks. Imaging agent for PSMA PET/CT.
  Other Names: 68Ga-PSMA-HBED-CC

SUMMARY:
This is a phase I/II dose-escalation study of 225Ac-J591 administered together with 177Lu-PSMA-I&T (also known as PNT2002). The two study drugs are 225Ac-J591 and 177Lu-PSMA-I&T. Both drugs are designed to deliver radiation to prostate cancer cells; they are known as radionuclide conjugates (radiation linked to antibodies/molecules that recognize prostate cancer cells). The first phase of the study (phase I) will determine the highest dose of the study drug that can be safely given. The second phase of the study (phase II) will determine the effectiveness of the drug combination in patients with prostate cancer.

DETAILED DESCRIPTION:
This clinical trial is for men with progressive metastatic castration-resistant prostate cancer (mCRPC). The two primary objectives of this trial are to determine the highest dose of 225Ac-J591 and 177Lu-PSMA-I&T that can be administered together (also known as maximum tolerated dose) with the recommended phase II dose and to determine the effectiveness of the drug combination. Patients who choose to participate in this study will have a screening visit to determine whether or not they are eligible for the study. Subject(s) enrollment will be done as 3+3 study design at each dose level. Initially at least 2 subject(s) will be enrolled in Cohort 1 and will receive 225Ac-J591 30 KBq (0.81 µCi) / kg plus 177Lu-PSMA-I&T 6.8 GBq (184 mCi) with dose escalation. The enrollment ceiling of the dose escalation portion of the study is up to 18 treated study participants (up to three groups, up to 6 at each dose level).177Lu-PSMA-I&T will be given at a fixed dose of 6.8 GBq. 225Ac-J591 will be given starting at 30 KBq/kg, with a subsequent dose-escalation by an increment of 5-10 KBq/kg to 40 KBq/kg. The two drugs will be co-administered every 8 weeks, for 2 cycles. Once the recommended phase II dose has been established, the phase II component will enroll up to 24 patients to further test efficacy.

Preliminary results of our trials of single-agent 225Ac-J591 (single dose, fractionated dose, multiple dose regimens point towards a dose-response relationship as well as dose-toxicity relationship. In our published trials of 177Lu-J591, a very small difference in administered radioactivity has been associated with large differences in efficacy (PSA response and overall survival) [Tagawa et al. 2013; Tagawa et al. 2019]. In addition, guidance by the FDA recommends more precise testing of radioactivity doses. Therefore, we plan to enroll an additional cohort "1.5" to be treated with 35 KBq/Kg to determine RP2D for this population of patients.

The primary efficacy measure will be proportion of patients with PSA decline and proportion of patients with 50%+ PSA decline. Other objectives include to determine the radiographic response rate, biochemical progression-free survival, and overall survival. During the study, patients will be closely monitored for adverse events (side effects); weekly x4 weeks, then every 2 weeks until completion of therapy, then every 4 weeks until patients start another therapy. Long-term follow-up will be every 6 months, for 3 years. During the phase I component, the adverse event assessment phase will be a minimum of 8 weeks after the last dose of 225Ac-J591 and 177Lu-PSMA-I&T. At screening, week 12, and week 24, patients will undergo imaging. Imaging will include 68Ga-PSMA-11 PET/CT. 68Ga-PSMA-11 is comprised of gallium-68, a radiotracer, linked to PSMA-11, a molecule that binds to PSMA. Patients with PSMA-positive tumors are eligible for the study. Additional imaging includes SPECT imaging on day 8 of each cycle, to evaluate radiation uptake into the tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of prostate
* Documented progressive metastatic CRPC based on Prostate Cancer Working Group 3 (PCWG3) criteria, which includes at least one of the following criteria: PSA progression, Objective radiographic progression in soft tissue, New bone lesions
* ECOG performance status of 0-2
* Have serum testosterone < 50 ng/dL. Subjects must continue primary androgen deprivation with an LHRH/GnRH analogue (agonist/antagonist) if they have not undergone bilateral orchiectomy
* Have previously been treated with at least one of the following: Androgen receptor signaling inhibitor (such as enzalutamide), CYP 17 inhibitor (such as abiraterone acetate)
* Have previously received taxane chemotherapy, been determined to be ineligible for taxane chemotherapy by their physician or refused taxane chemotherapy
* Age > 18 years
* Patients must have normal organ and marrow function as defined below: Absolute neutrophil count: >2,000 cells/mm3, Hemoglobin: ≥9 g/dL, Platelet count: >150,000 x 109/uL, Serum creatinine: <1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min/1.73 m2 by Cockcroft-Gault, Serum total bilirubin: <1.5 x ULN (unless due to Gilbert's syndrome in which case direct bilirubin must be normal), Serum AST and ALT: <1.5 x ULN in the absence of liver metastases; <3 x ULN if due to liver metastases (in both circumstances bilirubin must meet entry criteria)
* Ability to understand, and the willingness to sign, a written informed consent document

Exclusion Criteria:

* Implantation of investigational medical device ≤4 weeks of Treatment visit #1 (Day 1) or current enrollment in oncologic investigational drug or device study
* Use of investigational drugs ≤4 weeks or <5 half-lives of Treatment visit # 1(Day 1) or current enrollment in investigational oncology drug or device study
* Prior systemic beta-emitting bone-seeking radioisotopes. Prior radium-223 is allowed provided at least 90 days have lapsed since last dose
* Prior PSMA-targeted radionuclide therapy (prior PSMA-targeted isotopes used for imaging/diagnostic purposes are allowed, as is prior PSMA-targeted therapy that does not involve therapeutic radionuclides)
* Known active brain or leptomeningeal metastases
* History of deep vein thrombosis and/or pulmonary embolus within 1 month of Treatment visit #1
* Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
* Radiation therapy for treatment of PC ≤4 weeks of Treatment visit #1
* Patients on stable dose of bisphosphonates or denosumab, which have been started no less than 4 weeks prior to treatment start, may continue on this medication, however patients are not allowed to initiate bisphosphonate/Denosumab therapy during the DLT-assessment period of the study
* Having partners of childbearing potential and not willing to use a method of birth control deemed acceptable by the principle investigator and chairperson during the study and for at least 140 days after last study drug administration
* Currently active other malignancy other than non-melanoma skin cancer. Patients are considered not to have "currently active" malignancy if they have completed any necessary therapy and are considered by their physician to be at less than 30% risk of relapse
* Known history of myelodysplastic syndrome

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Metastatic Castrate Resistant Prostate Cancer
Enrollment: 48 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with dose limiting toxicity (DLT) of 225Ac-J591 and 177Lu-PSMA-I&T during dose-escalation phase. | Will be collected at the time of visit 1 through end of study or 100 months
  DLTs will be measured by utilizing the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Cumulative maximum tolerated dose (MTD) and recommended phase II dose 225Ac-J591 and 177Lu-PSMA I&T | Will be collected at the time of visit 1 through end of study or 100 months
  The dose that produces an "acceptable" level of toxicity or that, if exceeded, would put subjects at "unacceptable" risk for toxicity. Definition of the MTD usually relies on the sample, as MTD is defined as the dose level at which no more than one patient out of six experienced dose-limiting toxicity (DLT).
Proportion of PSMA+ subjects (by imaging criteria) with PSA decline following treatment with the combination of 225Ac-J591 and 177Lu-PSMA I&T. | Will be collected at the time of visit 1 through end of study or 100 months
  Proportion of patients achieving 50% or greater PSA decline (relative to baseline/pre-treatment PSA). Response may occur at any time following treatment initiation and prior to going off study or initiation of new therapy.

SECONDARY OUTCOMES:
Change in biochemical progression-free survival | Will be collected at the time of visit 1 through end of study or 100 months
  PSA progression will be defined as a rise of > 25% above either the pretreatment level or the nadir PSA level (whichever is lowest). PSA must increase by > 2 ng/ml to be considered progression.
Change in circulating tumor cells (CTC) count | Samples will be collected at screening, week 12, week 24.
  CTCs will be analyzed through blood specimen collection via CellSearch methodology lab testing
Number of subjects with radiographic response rate | Patients will undergo imaging at screening, week 12, and week 24.
  Response evaluation criteria in solid tumors RECIST (Version 1.1) criteria with prostate cancer working group 3 (PCWG3) modifications will be used.
Safety of treatment and adverse event rate | Will be collected at the time of visit 1 through end of study or 100 months.
  National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 is used to grade all adverse events
Overall survival following treatment with 225Ac-J591 and 177Lu-PSMA-I&T | Survival will be collected from Day 1 through study completion up to 100 months
  Overall survival will be captured through in-clinic or telephone contact with subjects
Change in disease assessment with 68Ga-PSMA-11 PET/CT prior to and following investigational treatment | Patients will undergo imaging at screening, week 12, and week 24.
  68Ga-PSMA-11 PET/CT will be utilized as part of the radiographic assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Osborne, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Brooklyn Methodist Hospital - New York Presbyterian, Brooklyn, New York
  - Weill Cornell Medicine New York Presbyterian, New York, New York

IPD SHARING:
Plan to Share IPD: No